CLINICAL TRIAL: NCT02116088
Title: Prevention and Intervention of Externalizing Problem Behavior in School: Development and Evaluation of a Teacher Coaching.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Collaborators: University of Applied Sciences Düsseldorf (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Manfred Doepfner, Univ. Prof. Dr., University of Cologne
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01JH1204B
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Problematic Behavior in Children
Keywords: Externalizing problem behavior, teacher training, teacher coaching, primary school, elementary school, continuing professional development, advanced training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receiving Teacher Coaching (Active Comparator): Teachers who currently take part in teacher coaching
  Interventions: Behavioral: Teacher Coaching
- Waiting for Teacher Coaching (No Intervention): Teachers who are currently waiting for taking part in teacher coaching

INTERVENTIONS:
Behavioral: Teacher Coaching
  Arms: Receiving Teacher Coaching

SUMMARY:
Children with externalizing problem behaviour are at risk of developing educational impairment, because of their problems in rule following, social behaviour and attention. This behaviour represents a great challenge for teacher. In addition, time pressures and conflicts with colleagues are the most common sources of stress for teachers. Till now teachers receive no evaluated training which in particular regards externalizing problem behaviour. Therefore we develop and evaluate an indicated prevention program for elementary school teachers with children with externalizing problem behaviour. All teachers of a participating school are given a general overview of externalizing problem behaviour (etiology, diagnosis) and information on evidence-based treatments for children with externalizing problem behaviour in school settings. Single teachers will then participate in a 12 week coaching in which they learn to apply classroom management techniques, strategies to improve their relationships with children, behaviour modification techniques and cognitive interventions to specific target children. The coaching intervention is based on functional behavioural analysis and provides teachers with evidence-based strategies which focuses on one target child.

Longitudinal data will be collected in a within-subject control group design. Dependent measures include teacher and observer reports.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 and 11 years, externalizing behavior problems

Exclusion Criteria:

-

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on Behavior in School Lessons (FVU) | one year

SECONDARY OUTCOMES:
Teacher´s Report Form (modified) | one year
Questionnaire on Attention Deficit Hyperactivity Disorder (FBB-ADHS) | one year
Questionnaire on Conduct Behavior Problems | one year
Brief Problem Monitor-Teacher Form (BPM-T/6-18) | one year
Weiss-Assessment Scale on Functional Impairment - Parent´s Report (WFIRS-P) | one year
Teacher Classroom Management Strategies Questionnaire (TSQ) | one year
Perceived Self-Efficacy of Teachers: Panel Design with a new Instrument (LSWS) | one year
The Index of Teaching Stress (ITS) | one year
Depression Anxiety Stress Scales (DASS) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Döpfner, Univ. Prof. Dr., Study Director — University Clinic of Cologne
Locations (1):
- University Clinic of Cologne, Cologne, North Rhine-Westphalia, Germany